CLINICAL TRIAL: NCT03806842
Title: Pivotal, Non-Randomized, Historically Controlled, Prospective, Multi-Center Clinical Study of the Easytech Reversed Shoulder System
Brief Title: Easytech Reversed Shoulder System Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: FX Shoulder Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FXUSA2018-01
Record Dates: First submitted 2018-12-31; First posted 2019-01-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Osteo Arthritis Shoulders; Avascular Necrosis of the Head of Humerus; Rotator Cuff Tear
Keywords: shoulder arthroplasty; reverse shoulder replacement
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: single arm, historically controlled, multi-center
Masking Description: no masking due to being a single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Easytech group (Other): patients who require a reverse total shoulder, meet the eligibility criteria and receive the Easytech Reversed Shoulder System
  Interventions: Device: Easytech group

INTERVENTIONS:
Device: Easytech group — total shoulder replacement

SUMMARY:
The purpose of the study is to collect data to demonstrate the safety and effectiveness of the Easytech Reversed Shoulder System for the treatment of patients who require a reverse total shoulder arthroplasty.

DETAILED DESCRIPTION:
The clinical study will enroll patient who require a reverse total shoulder arthroplasty as a result of osteoarthritis, post-traumatic arthritis, avascular necrosis and have a massive and non-repairable rotator cuff tear and a functional deltoid muscle.

If patients meet the eligibility criteria, evaluations and x-rays will be completed pre-operatively and post-operatively out to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are 21 years or older.
2. Patients are skeletally mature as evident by scapula and proximal humerus closure.
3. Patients exhibit clinical indications for primary reverse total shoulder arthroplasty based on physical exam and medical history including the following: osteoarthritis, post-traumatic arthritis, or avascular necrosis.
4. Patients have a massive and non-repairable rotator cuff tear.
5. Patients have a functional deltoid muscle.
6. Patients are anatomically and structurally suited to receive the implants;

   a. Subject show sufficient bone quality in the humerus bone intraoperatively via the thumb test, guide pin test, humeral punch test, and humeral anchor test as outlined in the surgical technique.
7. Patients with an adjusted Constant Score < 60 and ≥ 15.
8. Patients are willing and able to comply with the follow-up schedule and evaluation outlined in the protocol.
9. Patient are willing and able to sign the informed consent.

Exclusion Criteria:

1. Patients with Body Mass Index (BMI) greater than 40 kg/m2.
2. Patients have one of the following compromising the affected limb: a significant injury to the upper brachial plexus, paralysis of the axillary nerve or a neuromuscular disease compromising the affected limb which would render the procedure unjustifiable.
3. Patients have marked bone loss that would not allow sufficient support of the implant.
4. Patients have a known sensitivity or allergic reaction to one or more of the implanted materials.
5. Patients who are participating concurrently in another clinical study, or have participated in a clinical study within the last 90 days, or intend to during the course of the study.
6. Patients who have an active systemic infection, or an active local infection in or near the target shoulder, or have a previous history of joint infection.
7. Patients with known immunodeficiency.
8. Patients currently taking > 5mg/day corticosteroids (e.g. prednisone) excluding inhalers, within 3 months prior to surgery.
9. Patients with significant comorbidities as evident by an American Society of Anesthesiologists (ASA) score greater than 3.
10. Patients with active neoplastic disease.
11. Patients with current drug or alcohol abuse, or a history of the same within the last 6 months.
12. Patients with local circulatory problems, (e.g. thrombophlebitis and lymphedema).
13. Patients are pregnant or expect to become pregnant during the duration of the study.
14. Patients with any mental or psychological disorder that would impair their ability to complete the study questionnaires.
15. Patients with any medical condition or other circumstances that might interfere with their ability to return for follow-up visits in the judgment of the Investigator, including any systemic illness, neuromuscular, neurosensory, or musculoskeletal deficiency that would render the patient unable to perform appropriate postoperative rehabilitation.
16. Any condition which, in the judgment of the Investigator, would preclude adequate evaluation of device's safety and performance.
17. Patients with humeral or glenoid fractures.
18. Patients unable to stand from sitting position without the use of their hands/arms.
19. Patients with a history of fragility fractures as defined as any fall from a standing height or less, that results in a fracture.
20. Patients with osteoporosis, osteopenia, Paget's disease, osteomalacia or any other metabolic bone disease; a. Osteoporosis is defined as Simple Calculated Osteoporosis Risk Estimation (SCORE) above 6 and DXA (Dual-energy X-ray absorptiometry) T-score < -2.5 or QCT (Quantitative computed tomography) T-score < 80mg/cubic cm. History of a fragility fracture requires that a DXA scan or QCT scan is completed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Adjusted Constant-Murley Score | 24 months post-operative
  adjusted Constant Score of 70 or greater, no humeral radiolucency >2mm or humeral migration/subsidence >5mm, no revision surgery, no serious device related adverse event
no humeral radiolucency >2mm around the humeral component | 24 months post-operative
  on review of x-rays, there are no radiolucencies >2mm around the humeral component
no subsidence or migration of the humeral component >5mm | 24 months post-operative
  on review of x-rays, there is no subsidence or migration of the humeral component greater than or equal to 5mm
no revision | 24 months post-operative
  there is no revision of the humeral components
no serious device related adverse event | 24 months post-operative
  there is no serious device related adverse event reported

SECONDARY OUTCOMES:
QuickDASH | 24 months post-operative
  measures the ability to complete tasks, absorb forces and severity of symptoms
Visual Analog Scale for Pain (VAS) | 24 months post-operative
  on 100 point scale where 0 is no pain and 100 is severe pain
American Shoulder and Elbow Surgeon (ASES) | 24 months post-operative
  patient-reported outcomes with questions on function and pain
Range of Motion of the shoulder joint | 24 months
  forward and lateral elevation, internal & external rotation arm at side

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Trier, PhD, Study Director — FX Shoulder Solutions; Brian Rogers, BS, Study Director — FX Shoulder Solutions
Locations (6):
- United States (6):
  - The CORE Institute, Sun City West, Arizona
  - Dearborn & Associates Institute for Joint Reconstruction, Menlo Park, California
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Orthopedics Rhode Island, Wakefield, Rhode Island
  - Texas Orthopedic Specialists, Bedford, Texas
  - Carrell Clinic, Dallas, Texas

REFERENCES:
- See also: Company website — http://fxshouldersolutions.com